CLINICAL TRIAL: NCT02234986
Title: A Phase 2, Multi-center, Open-label Study of Oral ENMD-2076 for the Treatment of Patients With Advanced Fibrolamellar Carcinoma (FLC)
Brief Title: A Multi-center, Open-label Study of Oral ENMD-2076 for the Treatment of Patients With Advanced Fibrolamellar Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2076-CL-006
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; Advanced Fibrolamellar Carcinoma
Keywords: Advanced Fibrolamellar Carcinoma
MeSH Terms: interventions — ENMD 2076

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENMD-2076 (Experimental): ENMD-2076, oral capsule Once daily dose 250 mg/day
  Interventions: Drug: ENMD-2076

INTERVENTIONS:
Drug: ENMD-2076 — 250 mg oral dose, once daily (QD) for 28 day cycles

SUMMARY:
The purpose of the study is to determine whether once-daily dosing with ENMD-2076 will be a safe and effective treatment in patients with FLC. Safety will be measured by looking at the adverse events that may happen and the efficacy will look at the progression of the disease over time.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the 6-month progression free survival (PFS6) rate when patients with advanced fibrolamellar carcinoma (FLC) are treated with daily oral ENMD 2076

Secondary Objectives:

* To evaluate the overall response rate using RECIST v 1.1 criteria when patients with FLC are treated with daily oral ENMD 2076.
* To evaluate the median Progression Free Survival (PFS), Time to Progression (TTP), and Overall Survival (OS).
* To determine the safety of ENMD-2076 as defined by the frequency and severity of adverse events when patients with FLC are treated with daily oral ENMD-2076

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced fibrolamellar carcinoma (FLC).
* All forms of prior local therapy are allowed as long as patients have either a target lesion, which has not been treated with local therapy and/or the target lesion(s) within the field of the local-regional therapy has shown an increase of ≥ 20% in size. Local-regional therapy must be completed at least 4 weeks prior to the baseline CT scan. Local therapies including chemoembolization do not count as prior systemic therapy.
* Are at least 4 weeks from major surgery and recovered.
* At least one measureable lesion by RECIST 1.1.
* Male or non-pregnant, non-breastfeeding female at least 18 years of age. Patients aged at 12~18 years may be recruited but only at the site principle investigator's request and subject to Institutional Review Board (IRB) approval.
* Has a pre-study echocardiogram or multi-gated acquisition (MUGA) scan with an actual left ventricular ejection fraction of greater than or equal to the institutional lower limit of normal within one month of initiating therapy.
* Have clinically acceptable laboratory screening results within certain limits specified below:

  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times upper limit of normal (ULN)
  * Total bilirubin ≤ 3.0 x ULN
  * Creatinine ≤ 1.5 x ULN or Cr Cl > 60 cc/min
  * Absolute neutrophil count ≥ 1500 cells/mm3
  * Platelets ≥ 50,000/mm3
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 for ≥ 16 years of age and a Lansky performance status of 70-100 for < 16 years of age
* Women and men of child producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication. A serum pregnancy test within 72 hours prior to the initiation of therapy will be required for women of childbearing potential.
* Have the ability to understand the requirements of the study, provide written informed consent, which includes authorization for release of protected health information, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

* Have active, acute, or chronic clinically significant infections or bleeding within the last 6 months or previous thromboembolic or hemorrhagic events during anti angiogenic therapy.
* Have uncontrolled hypertension (systolic blood pressure greater than 150 or diastolic blood pressure greater than 100) or history of congestive heart failure (AHA Grade 2 or higher).
* Have active angina pectoris, stroke or recent myocardial infarction (within 6 months).
* Have uncontrolled chronic atrial fibrillation.
* Have chronic atrial fibrillation or QTc interval corrected for heart rate of greater than 470 msec in adults and 450 msec in pediatrics (< 18 years).
* Have additional uncontrolled serious medical or psychiatric illness that in the point of view of the investigator can render the patient unable to receive therapy or make it unsafe to receive therapy.
* Require treatment with any of the exclusionary medications listed in Appendix D.
* Known untreated or unstable central nervous system (CNS) metastatic disease.
* Have persistent 2+ protein by urinalysis (patients with 2+ proteinuria that have a spot protein:creatinine ratio of less than 0.3 may be enrolled) or a history of nephrotic syndrome.
* Subjects with history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the investigator will not affect patient outcome in the setting of current FLC diagnosis.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Ren, PhD, Study Director — CASI Pharmaceuticals, Inc.; Ghassan Abou-Alfa, MD, Study Chair — MSKCC
Locations (5):
- United States (5):
  - CASI Site 03, San Francisco, California
  - CASI Site 04, Aurora, Colorado
  - CASI Site 02, Boston, Massachusetts
  - Casi Site 01, New York, New York
  - CASI Site 05, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abou-Alfa GK, Mayer R, Venook AP, O'Neill AF, Beg MS, LaQuaglia M, Kingham PT, Kobos R, Basturk O, Brennan C, Yopp A, Harding JJ, Leong S, Crown J, Hoti E, Leonard G, Ly M, Bradley M, Valentino E, Markowitz D, Zukiwski A, Ren K, Gordan JD. Phase II Multicenter, Open-Label Study of Oral ENMD-2076 for the Treatment of Patients with Advanced Fibrolamellar Carcinoma. Oncologist. 2020 Dec;25(12):e1837-e1845. doi: 10.1634/theoncologist.2020-0093. Epub 2020 Mar 10. PMID 32154962

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 patients screened; 35 patients enrolled
Period: Overall Study
Arm/Group | ENMD-2076
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 35 patients were enrolled; all patients were evaluable for toxicity and efficacy
Groups:
- ENMD-2076: ENMD-2076, oral capsule Once daily dose 250 mg/day 28 day cycles
Arm/Group | ENMD-2076
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 25 [12 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Eastern Cooperative Oncology Group (ECOG) status [Number; unit: participants] — ECOG status was applicable to patients with age >= 16 years. Population: 33 of the 35 patients in this study was >= 16 years of age.
  participants
    ECOG 0: Fully active, able to carry on all pre-disease performance without restriction: number analyzed (Participants) | 33
    ECOG 0: Fully active, able to carry on all pre-disease performance without restriction | 12
    ECOG 1: Restricted in physically strenuous activity but ambulatory, able do work of a light nature: number analyzed (Participants) | 33
    ECOG 1: Restricted in physically strenuous activity but ambulatory, able do work of a light nature | 19
    ECOG 2: Ambulatory and capable of selfcare, unable to carry out any work; up >50% of waking hours: number analyzed (Participants) | 33
    ECOG 2: Ambulatory and capable of selfcare, unable to carry out any work; up >50% of waking hours | 2
Lansky status [Number; unit: participants] — Only applied to patients <16 years of age. Population: Lansky status was applicable to patients < 16 years of age. Two patients enrolled in the study were < 16 years of age.
  participants
    Lansky 100: Fully active: number analyzed (Participants) | 2
    Lansky 100: Fully active | 1
    Lansky 90: Minor restriction in physically strenuous play: number analyzed (Participants) | 2
    Lansky 90: Minor restriction in physically strenuous play | 1
Number of prior systemic therapies [Median (Full Range); unit: Number of prior systemic therapies] | 4 [3 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: 6-month overall response rate (ORR rate) using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR) - disappearance of all target lesions; partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; ORR = proportion of patients evaluated as CR + PR
Time Frame: 6 months
Population: Patients treated and evaluable for efficacy
Measure: Count of Participants; unit: Participants
Groups:
- ENMD-2076: ENMD-2076, oral capsule Once daily dose 250 mg/day
  ENMD-2076: 250 mg oral dose, QD for 28 day cycles
Arm/Group | ENMD-2076
Number analyzed (Participants) | 35
Participants
  Partial response | 1
  Stable disease | 20
  Progressive disease | 10
  Other / unknown | 4

2. Secondary Outcome: Progression Free Survival
Description: using RECIST v 1.1 criteria
Time Frame: 6 months
Population: patients treated and evaluable for efficacy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ENMD-2076
Number analyzed (Participants) | 35
months | 3.9 [2.3 to 5.5]

3. Other Pre Specified Outcome: Frequency and Severity of Adverse Events
Description: Frequency and severity of adverse events in patients evaluable for toxicity
Time Frame: 6 months
Population: patients treated and evaluable for toxicity assessment; regardless of relationship to study medication according to CTCAE 5.0
Measure: Count of Participants; unit: Participants
Arm/Group | ENMD-2076
Number analyzed (Participants) | 35
Participants
  Fatigue | 27
  ALT increased | 26
  AST increased | 24
  Abdominal pain | 23
  Diarrhea | 23

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | ENMD-2076
All-Cause Mortality (participants affected / at risk) | 3/35
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENMD-2076 (N=35)
Sepsis (Infections and infestations) | 1 (1) — unlikely related to study drug
Liver failure (Hepatobiliary disorders) | 1 (1) — possibly related to study drug
Respiratory failure (Cardiac disorders) | 1 (1) — unlikely related to study drug
Seizure (Nervous system disorders) | 1 (1) — possibly related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENMD-2076 (N=35)
Fatigue (General disorders) | 27 (27)
Fever (General disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 20 (20)
Vomiting (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 23 (23)
Constipation (Gastrointestinal disorders) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Decreased neutrophil count (Blood and lymphatic system disorders) | 2 (2)
Decreased platelet count (Investigations) | 5 (5)
Increased hemoglobin (Investigations) | 4 (4)
INR increased (Investigations) | 3 (3)
Prolonged aPTT (Investigations) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Weight loss (Investigations) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (10)
Hypertension (Vascular disorders) | 16 (16)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 24 (24)
Abdominal pain (Gastrointestinal disorders) | 23 (23)
Alanine aminotransferase increased (Investigations) | 26 (26)
Alkaline phosphatase increased (Investigations) | 15 (15)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (17)
Hyponatremia (Metabolism and nutrition disorders) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Headache (Nervous system disorders) | 12 (12)
Insomnia (Psychiatric disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Proteinuria (Renal and urinary disorders) | 7 (7)
Blurred vision (Eye disorders) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Encephalopathy (Nervous system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Blood bilirubin increased (Investigations) | 6 (6)
Non-cardiac chest pain (General disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 3 (3)
Enteritis (Infections and infestations) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Pain (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT02234986/Prot_SAP_000.pdf